CLINICAL TRIAL: NCT06836934
Title: SOFT KNEE BRACE VERSUS LATERAL WEDGE FOOT INSOLE on PAIN and PROPRIOCEPTION in KNEE OSTEOARTHRITIS PATIENTS.
Brief Title: Soft Knee Brace Versus Lateral Wedge in Knee Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, omar hashem abd el moamen elsayed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005582
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthristis
Keywords: knee osteoarthritis soft knee brace lateral wedge foot insole; proprioception pain

STUDY DESIGN:
Intervention Model Description: soft knee brace and lateral wedge foot insole
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- conventional physical therapy (Active Comparator): the patient will receive treatment For 8weeks three times a week
  Strengthening Exercises:
  * Quadriceps Strengthening: Exercises like straight leg raises, quadriceps sets, and seated knee extensions help strengthen the quadriceps muscle, which supports the knee joint.
  * Hamstring Strengthening: Hamstring curls and bridges target the hamstrings to enhance stability and support for the knee.
  * Hip Strengthening: Exercises such as hip abductions, adductions, and clamshells strengthen the hip muscles (each 3 sets, 10 reps).
  Flexibility Exercises:
  * Hamstring Stretch: Gentle stretching of the hamstrings can alleviate tension around the knee.
  * Quadriceps Stretch: Stretches like the standing quadriceps stretch help maintain flexibility in the front of the thigh.
  * Calf Stretch: Stretching the calf muscles can prevent tightness TENS (Transcutaneous Electrical Nerve Stimulation): Helps manage pain by sending electrical impulses to the affected area.
  Interventions: Procedure: convential physical therapy program
- soft knee brace (Experimental): the patient will Wear soft knee brace for 8 weeks plus traditional physical therapy A commercially available soft brace (orthopedics ser. number 86) plus traditional physiotherapy The patient will wear the brace brace except for sleeping
  A tight brace was defined as one that was fitted based on shank and thigh circumferences measured according to instructions provided by the distributor (standard fit). A non-tight brace was defined as being 1 size larger than a tight brace. plus conventional therapy Strengthening Exercises:
  * Quadriceps Strengthening: Exercises like straight leg raises, quadriceps sets, and seated knee extensions help strengthen the quadriceps muscle, which supports the knee joint.
  * Hamstring Strengthening: Hamstring curls and bridges target the hamstrings to enhance stability and support for the knee.
  * Hip Strengthening: Exercises such as hip abductions, adductions, and clamshells strengthen the hip muscles (each 3 sets, 10 reps). (Deyle et al ., 2005) Flexibil
  Interventions: Device: soft knee brace; Procedure: convential physical therapy program
- lateral wedge foot insole (Experimental): the patient will wear Lateral wedge insole 5mm for 8 weeks plus traditional physical therapy
  Standardized non-customized laterally wedged insoles were evaluated. Insoles were made of high-density ethyl vinyl acetate, were wedged approximately 5° (as greater wedging is associated with foot discomfort and were worn inside the participant's own shoes. In loaded positions ,The insoles were wedged along the lateral edge of the entire length of the foot. Strengthening Exercises:
  * Quadriceps Strengthening: Exercises like straight leg raises, quadriceps sets, and seated knee extensions help strengthen the quadriceps muscle, which supports the knee joint.
  * Hamstring Strengthening: Hamstring curls and bridges target the hamstrings to enhance stability and support for the knee.
  * Hip Strengthening: Exercises such as hip abductions, adductions, and clamshells strengthen the hip muscles (each 3 sets, 10 reps). (Deyle et al ., 2005)
  Flexibility Exercises:
  • Hamstring Stretch: Gentle stretc
  Interventions: Device: lateral wedge foot insole; Procedure: convential physical therapy program

INTERVENTIONS:
Device: soft knee brace — A commercially available soft brace (orthomedics ser. number 86) plus traditional physiotherapy
  Arms: soft knee brace
Device: lateral wedge foot insole — Wearing Lateral wedge insole 5mm for 8 weeks Standardized non-customized laterally wedged insoles were evaluated. Insoles were made of high-density ethyl vinyl acetate, were wedged approximately 5°
  Arms: lateral wedge foot insole
Procedure: convential physical therapy program — Strengthening Exercises:
  * Quadriceps Strengthening: Exercises like straight leg raises, quadriceps sets, and seated knee extensions help strengthen the quadriceps muscle, which supports the knee joint.
  * Hamstring Strengthening: Hamstring curls and bridges target the hamstrings to enhance stability and support for the knee.
  * Hip Strengthening: Exercises such as hip abductions, adductions, and clamshells strengthen the hip muscles (each 3 sets, 10 reps). (Deyle et al ., 2005)
  Flexibility Exercises:
  * Hamstring Stretch: Gentle stretching of the hamstrings can alleviate tension around the knee.
  * Quadriceps Stretch: Stretches like the standing quadriceps stretch help maintain flexibility in the front of the thigh.
  * Calf Stretch: Stretching the calf muscles can prevent tightness (J. D. Deyle et al 2005) TENS (Transcutaneous Electrical Nerve Stimulation): Helps manage pain by sending electrical impulses to the affected area.

SUMMARY:
the aim of study is to investigate the efficacy of soft knee brace versus lateral wedge foot insole on pain and proprioception in knee OA

DETAILED DESCRIPTION:
Osteoarthritis is the most common disease of joints in adults around the world. Felson et al. reported that about one-third of all adults have radiological signs of osteoarthritis.

. according to epidemiological study the prevalence of knee osteoarthritis in the The Middle East and North Africa ( MENA) region increased 2.88-fold, from 6.16 million cases to 17.75 million, between 1990 and 2019 in MENA.

Individuals with knee OA may have a variety of impairments and functional limitations that prevent them from participating in regular exercise and physical activity. Physical therapists can offer a variety of supplemental treatment approaches that may help patients overcome these barriers and enhance the overall effectiveness of exercise therapy programs.

Soft braces are elastic, non-adhesive orthoses recommended in the non-surgical management of patients with knee osteoarthritis (OA). Because of ease of use, lack of complications, and low cost, soft braces are commonly used with the aim of reducing pain and activity limitations.

.according to Cudejko ,study in 2019 This study shows that decreased pain and reduced dynamic knee instability are pathways by which wearing a soft knee brace decreases activity limitations in patients with knee OA.

Osteoarthritis wedged insoles for patients with medial compartment knee osteoarthritis is certainly a very interesting treatment option because of its low cost, low complexity and virtually absence of side effects.

To reduce pain, improve physical function, and, possibly, slow disease progression in KOA, the use of knee braces has often been suggested. These are generally the main purposes of knee braces, but the optimal choice for an orthosis remains unclear, and long-term implications are lacking. A variety of different bracing types, manufacturers, and products are currently available on the market. Short-lever elastic knee braces have been used to improve pain, specifically during squats or walking, and daily use or the use of soft knee braces while resting is suggested to provide moderate pain relief and small-to-moderate effects on performance-based physical function in patients. Several authors, with respect to these findings, highlight the importance of soft braces to improve pain reduction and physical function in both the short and long term in KOA treatment, but additional high-quality studies are warranted to improve confidence in the findings

that lateral wedge insoles may be modestly effective in reducing pain in patients with medial knee OA. However, the treatment effect was small and most treated patients did not achieve conventional levels of min imally important response. Future modifications of the screening strategy or treatment might offer greater levels of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Their ages range from 40-60 years old.
2. The patients included to this study according to American College of Rheumatology (ACR) criteria, namely, knee pain; and/or morning stiffness longer than 30 minutes and/or joint crepitus.
3. The patients Kellgren Lawrence scores grade II-IV.
4. All the patients included had a minimum score of 25 on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total scores.
5. Unilateral symptomatic knee.

Exclusion Criteria:

* 1. high tibial osteotomy other realignment surgery 2. knee replacement 3. knee arthroscopy within the last 6 months. 4. an intraarticular injection within the past 3 months. 5. rheumatoid arthritis or patellofemoral syndrome 6. diabetic neuropathic pain or fibromyalgia. 7. foot or ankle problems that contraindicated the use of load-modifying interventions in footwear 8. body mass index (BMI) ≥35 kg/m2.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-02-26 (Estimated)

PRIMARY OUTCOMES:
pain intenisty | 2 months
  The visual analog scale (VAS) is the VAS, which consists of a line, usually 10 cm long, ranging from no pain or discomfort (zero) to the worst pain that could possibly feel (10)

SECONDARY OUTCOMES:
proprioception | 2 months
  Digital inclinometer is a valid tool alternative for isokinetic dynamometer in measuring active knee JPS in OA individuals at target angle 30˚ of knee flexion. However, there were high intra-class reliability and low inter-class reliability at target angle 30˚ of knee flexion. Also, the study revealed that another type of digital inclinometer (SPI Tronic, Penn tool co, Maplewood, NJ) is reliable and valid
physical function | 2 months
  The WOMAC Osteoarthritis Index(English version) has been assessed for validity and reliability and it was reports that it is valid and reliable .The original English language version of the WOMAC Osteoarthritis Index has been translated and validated into more than fifty languages as German(7), French(8), Spanish(9), Italian (10), Turkish(11), Moroccan (12) and classic Arabic(13).The classic Arabic version of the WOMAC(ArWOMAC) was in literal Arabic language to match the largest Arab population use.
range of motion | 2 months
  Knee flexion ROM measurement The individual was placed at dorsal decubitus, with 90 degrees of hip flexion. Hip positioning was guaranteed using a thigh device which aided in the maintenance of the pre-set position.
  The digital inclinometer was placed proximally and anteriorly on the leg, resting on the tibial crest.
  Knee extension ROM measurement The individual was at dorsal decubitus, with extended legs. The evaluated limb was raised by the heel, with knee stabilization in contact with the stretcher. The instruments positioning in relation to the segment was the same as the measurements performed for knee flexion.

CONTACTS AND LOCATIONS:
Overall Officials: omar ha abdelmoamen el sayed, Principal Investigator — cairo universty
Locations (1):
- Cairo Universty, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided